CLINICAL TRIAL: NCT01537432
Title: Phase II Randomized Double Blinded Placebo Controlled, Multiple-dose Regimen Study to Assess the Rate of Histological Clearance and Effect on Molecular Pathways as Well as on Biomarkers of 12 Months Secukinumab 300 mg s.c. Treated Patients With Chronic Plaque-type Psoriasis
Brief Title: Multiple-dose Regimen Study to Assess Effect of 12 Months of Secukinumab Treatment on Skin Response and Biomarkers in Psoriasis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A2223
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Results first posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-11

CONDITIONS: Psoriasis, Plaque-type Psoriasis
Keywords: Psoriasis, Plaque-type psoriasis; Plaque; Secukinumab; AIN457A; PASI; DLQI; IGA
MeSH Terms: conditions — Psoriasis; Plaque, Amyloid | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo
- secukinumab (Experimental): secukinumab
  Interventions: Drug: secukinumab

INTERVENTIONS:
Drug: secukinumab — secukinumab
  Arms: secukinumab
Drug: placebo — placebo comparator
  Arms: placebo

SUMMARY:
This study is designed to evaluate the proportion of patients achieving reversal of chronic plaque psoriasis at week 4 and 12 following multiple doses of secukinumab administered subcutaneously (sc) compared to placebo. Starting from week 13, all patients will receive multiple doses of secukinumab up to week 52 to study long term effects of secukinumab. Clinical endpoints including biomarker assessments, PASI, IGA and DLQI will be compared to better understand, why secukinumab may be effective in psoriasis patients.

ELIGIBILITY:
Inclusion criteria:

* Chronic plaque-type psoriasis diagnosed for at least 6 months
* Moderate to severe psoriasis as defined by: PASI score of ≥12, IGA score of ≥3, BSA (body surface area) affected by plaque-type psoriasis of ≥10%
* Chronic plaque-type psoriasis considered inadequately controlled by: topical treatment and/or; phototherapy and/or previous systemic therapy

Exclusion criteria:

* Forms of psoriasis other than chronic plaque-type
* Evidence of skin conditions at the time of the screening visit (e.g., eczema) that would interfere with evaluations of the effect of the investigational product on psoriasis
* History or evidence of active tuberculosis or evidence of latent tuberculosis (or other infections like Hepatitis-C/B), malignancy; active or known use of other immunosuppressive drugs (for eg: AIDs, RA, organ rejection etc.) at the screening visit
* Pregnant or nursing (lactating) women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (12):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, East Windsor, New Jersey
  - Novartis Investigative Site, Verona, New Jersey
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- AIN457 300mg: AIN457 300mg subcutaneously weekly
- Placebo: Placebo subcutaneously weekly until Week 12. At week 12, participants received AIN457 300mg subcutaneously weekly.
Period: Overall Study
Arm/Group | AIN457 300mg | Placebo
Started | 24 | 12
Completed | 18 | 10
Not Completed | 6 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Administrative problems | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Unsatisfactory therapeutic effect | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 300mg | Placebo | Total
Number analyzed (Participants) | 24 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (14.0) | 50.3 (13.8) | 48.4 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 17 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Skin Histology Response After Secukinumab Treatment From Baseline to Week 12
Description: Histological sections of lesional and nonlesional skin biopsies at baseline and at Week 12 were examined. For each visit, each patient's lesional skin biopsy was scored for the degree of histological improvement compared to that patient's baseline disease on a five point scale; -
  1 (worse) to +3 (excellent). Histological disease reversal or "excellent improvement" (histological disease reversal score = 3) was declared at the endpoint when all of the following four criteria were met.
Time Frame: Baseline, Week 12
Population: PharmacoDynamic PD -All patients with at least one evaluable post-treatment PD measurement and no protocol deviations with relevant impact on PD data.
Measure: Number; unit: percentage of participants
Arm/Group | AIN457 300mg | Placebo
Number analyzed (Participants) | 23 | 12
percentage of participants | 56.5 | 0.0
Statistical Analysis 1: Comparison: AIN457 300mg vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact; difference in proportions = 0.565, 95% CI 2-sided [0.363 to 0.768]

2. Secondary Outcome: Percentage of Participants Achieving Skin Histological Disease Reversal at Week 52
Description: Histological sections of lesional and nonlesional skin biopsies at Week 52 were examined. For each visit, each patient's lesional skin biopsy was scored for the degree of histological improvement compared to that patient's baseline disease on a five point scale; -
  1 (worse) to +3 (excellent). Histological disease reversal or "excellent improvement" (histological disease reversal score = 3) was declared at the endpoint when all of the following four criteria were met.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | AIN457 300mg | Placebo
Number analyzed (Participants) | 24 | 12
percentage of participants | 62.5 | 33.3

ADVERSE EVENTS:
Groups:
- AIN457 300 mg: AIN457 300mg subcutaneously weekly
Arm/Group | AIN457 300 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/12
Other Adverse Events (participants affected / at risk) | 13/24 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300 mg (N=24) | Placebo (N=12)
Lobar pneumonia (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300 mg (N=24) | Placebo (N=12)
Ear pain (Ear and labyrinth disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Fatigue (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 5 | 3
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Weight increased (Investigations) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.